CLINICAL TRIAL: NCT04788888
Title: VANTAGE Clinical Trial Evaluation of TAVR Using the NAVITOR Valve in a Global Investigation
Brief Title: Evaluation of TAVR Using the NAVITOR Valve in a Global Investigation
Acronym: VANTAGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10342
Record Dates: First submitted 2021-03-02; First posted 2021-03-09 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Symptomatic Severe Aortic Stenosis
Keywords: NAVITOR Heart disease; Transcatheter aortic valve implantation (TAVI); Aortic stenosis Cardiovascular disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Navitor Transcatheter Aortic Valve, FlexNav Delivery System (Experimental): Navitor Transcatheter Aortic Valve System Navitor valves (23mm, 25mm, 27mm, 29mm, and 35mm Titan valve), FlexNav Delivery system (small and large) and and Navitor Loading System (small, large, and LG+)
  Interventions: Device: Navitor Transcatheter Aortic Valve and FlexNav Delivery System

INTERVENTIONS:
Device: Navitor Transcatheter Aortic Valve and FlexNav Delivery System — For traditional application, the Navitor valve is indicated for transcatheter delivery in patients with symptomatic severe native aortic stenosis who are intermediate or low surgical risk.
  For the valve-in-valve application, the Navitor valve is indicated for use in patients with symptomatic heart disease due to failure (stenosed, insufficient, or combined) of a surgical bioprosthetic aortic valve.
  Subjects will undergo transcatheter aortic valve replacement (TAVR) with the Navitor valve and FlexNav Delivery system

SUMMARY:
Evaluation of TAVR using the NAVITOR valve in a Global Investigation.

DETAILED DESCRIPTION:
The VANTAGE clinical trial will evaluate the safety and effectiveness of the Navitor valve in patients with severe, symptomatic aortic stenosis who are at intermediate or low risk of surgical mortality. This trial will also evaluate the safety and effectiveness of the Navitor valve in a valve-in-valve application.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who is judged by a Heart Team, including a cardiac surgeon, to be appropriate for transcatheter heart valve intervention therapy, and is deemed to be at intermediate or low risk for open surgical aortic valve replacement (i.e., heart team estimates risk of surgical mortality < 7% at 30 days, considering the Society of Thoracic Surgeons (STS) risk score, overall clinical status, and other clinical co-morbidities unmeasured by the risk calculator). *
2. New York Heart Association (NYHA) Functional Classification of II, III, or IV *
3. Degenerative aortic valve stenosis with echo-derived criteria, defined as:

   aortic valve area (AVA) of ≤ 1.0 cm2 (or indexed EOA ≤ 0.6 cm2/m2) AND either mean gradient ≥ 40 mmHg or peak jet velocity ≥ 4.0 m/s or doppler velocity index (DVI) ≤ 0.25. The echocardiogram supporting the qualifying AVA baseline measurement must be performed within 90 days prior to informed consent). *
4. Aortic annulus diameter of 19-30 mm and ascending aorta diameter of 26-44 mm for the specified valve size listed in the IFU, as measured by CT (systolic phase) conducted within 12 months prior to informed consent.

Exclusion Criteria:

1. Life expectancy is less than 2 years in the opinion of the Investigator.
2. Evidence of an acute myocardial infarction [defined as ST-segment elevation myocardial infarction (STEMI) or non-ST-segment elevation myocardial infarction (NSTEMI) with acute ischemia symptoms and troponin elevation] within 30 days prior to index procedure.
3. Untreated clinically significant coronary artery disease requiring revascularization.
4. Any percutaneous coronary or peripheral interventional procedure performed within 30 days prior (except pacemaker or implantable cardioverter defibrillator (ICD) implant) to index procedure or planned within 30 days following the index procedure.
5. Blood dyscrasias as defined: leukopenia (WBC < 3000 mm3), acute anemia (Hb < 9 g/dL), thrombocytopenia (platelet count < 50,000 cells/mm³); history of bleeding diathesis or coagulopathy
6. Active peptic ulcer or upper GI bleeding within 3 months prior to index procedure that would preclude anticoagulation
7. Recent (within 6 months prior to index procedure date) cerebrovascular accident (CVA) or a transient ischemic attack (TIA)
8. Renal insufficiency (creatinine > 3.0 mg/dL or eGFR < 30 ml/min/1.73m2) and/ or end stage renal disease requiring chronic dialysis
9. Hostile chest or conditions or complications from prior surgery that would make the subject be considered high surgical risk (i.e., mediastinitis, radiation damage, abnormal chest wall, porcelain aorta, adhesion of aorta or internal mammary artery to sternum, etc.) *
10. Significant frailty as determined by the heart team (after objective assessment of frailty parameters) that would indicate high or extreme surgical risk *
11. Mixed aortic valve disease (aortic stenosis and aortic regurgitation with predominant aortic regurgitation 3-4+) *
12. Aortic valve is a congenital unicuspid or congenital bicuspid valve as verified by echocardiography or CT *
13. Severe ventricular dysfunction with LVEF < 30% as measured by resting echocardiogram
14. Pre-existing prosthetic heart valve or other implant (such as prosthetic ring or transcatheter edge-to-edge repair (TEER) clip) in any valve position * (Note: Subjects with a bioprosthetic aortic valve may be included in the ViV cohort.)
15. Severe circumferential mitral annular calcification (MAC) which is continuous with calcium in the left ventricular outflow tract (LVOT) *
16. Severe (greater than or equal to 3+) mitral regurgitation or severe mitral stenosis with pulmonary compromise
17. Minimum access vessel diameter of < 5.0 mm for small FlexNav Delivery System and < 5.5 mm for large FlexNav Delivery System
18. Eccentricity ratio of the annulus < 0.73

    * Criterion not applicable for valve-in-valve application

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Estimated)
Dates: Start 2021-06-13 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2036-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of a composite of all-cause mortality or fatal stroke/stroke with disability at 12 months (Primary Safety Endpoint) | 12 months post index procedure
  A composite of all-cause mortality or fatal stroke/stroke with disability at 12 months post index Navitor implantation procedure per the Valve Academic Research Consortium (VARC) 3 event definitions
The proportion of subjects who have moderate or greater paravalvular leak at 30 days (Primary Effectiveness Endpoint) | 30 days post index procedure
  Moderate or greater paravalvular leak at 30 days

SECONDARY OUTCOMES:
Transvalvular gradient | 12 months post index procedure
  Mean change in mean transvalvular gradient between baseline and 12 months
Effective orifice area | 12 months post index procedure
  Mean change in effective orifice area between baseline and 12 months
KCCQ quality of life score | 12 months post index procedure
  Mean change in KCCQ quality of life score between baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Worthley, M.D., Ph. D., Principal Investigator — Macquarie University Hospital; Nicolas van Mieghem, M.D., Ph. D., Principal Investigator — Erasmus Medical Center; Barathi Sethuraman, Study Director — Abbott
Locations (39):
- Australia (6):
  - St. Andrew's Hospital, Adelaide
  - The Alfred Hospital, Melbourne
  - Fiona Stanley Hospital, Murdoch
  - Macquirie University Hopsital, Ryde
  - Prince of Wales Hospital, Sydney
  - Princess Alexandra Hospital, Woolloongabba
- Austria (3):
  - Universitätsklinik Graz, Graz
  - Kepler Universitätsklinikum GmbH, Linz
  - AKH Wien, Vienna
- Rigshospitalet, Copenhagen, Denmark
- France (3):
  - CHU Gabriel Montpied, Clermont-Ferrand
  - Hopital Haut Leveque, Pessac
  - Clinique Pasteur Toulouse, Toulouse
- Germany (9):
  - Kerckhoff-Klinik GgmbH, Bad Nauheim
  - Universitätsmedizin Berlin - Charité Campus Mitte (CCM), Berlin
  - St. Johannes-Hospital, Dortmund
  - Herzzentrum Dresden, Dresden
  - Klinikum der Johann Wolfgang Goethe-Universität Frankfurt, Frankfurt
  - UKE Hamburg (Universitatsklinik Eppendorf), Hamburg
  - Herzzentrum Leipzig GmbH, Leipzig
  - Universität Mainz (Johannes Gutenberg-Universität Mainz), Mainz
  - DHZ München, München
- Shaare Zedek Medical Center, Jerusalem, Telaviv, Israel
- Italy (5):
  - Pineta Grande Hospital, Castel Volturno, Caserta
  - Azienda Ospedale Università Padova, Padua, Padua
  - Policlinico San Donato, Milan
  - Centro Cardiologico Monzino, Milan
  - Ospedale San Raffaele - Cardiac, Milan
- Erasmus MC - Thoraxcenter, Rotterdam, Netherlands
- Spain (5):
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Ramón y Cajal, Madrid
  - Hospital Clinico Universitario San Carlos, Madrid
  - Hospital Virgen de Rocio, Seville
- HerzZentrum Hirslanden, Zurich, Switzerland
- United Kingdom (4):
  - Royal Victoria Hospital, Belfast
  - Leeds General Infirmary, Leeds
  - Kings College Hospital, London
  - Morriston Hospital, Swansea

IPD SHARING:
Plan to Share IPD: No